CLINICAL TRIAL: NCT04855942
Title: Focused Extracorporeal Shock Wave Therapy (ESWT) Versus Traditional Physiotherapy in the Treatment of Trigger Finger: a Randomized Controlled Study
Brief Title: Focused Extracorporeal Shock Wave Therapy (ESWT) Versus Traditional Physiotherapy in the Treatment of Trigger Finger
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the outbreak COVID-19 in our country, the patients coming to our hospital drastically decreased. We could hardly enroll participants due to the paucity of our patients for more than six months, so we decided to withdrawn this study.
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (811)109A-50
Record Dates: First submitted 2021-03-10; First posted 2021-04-22 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Trigger Finger; Stenosing Tenosynovitis
Keywords: extracorporeal shock wave; trigger finger; stenosing tenosynovitis
MeSH Terms: conditions — Trigger Finger Disorder; Tendon Entrapment | interventions — Extracorporeal Shockwave Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Our study design is mainly to compare the therapeutic effect to trigger finger between extracorporeal shock wave (PiezoWave2 ECO, produced by Richard Wolf) and traditional physiotherapy.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Focused Extracorporeal Shock Wave Therapy (ESWT) (Experimental): 2000 impulses of 5 Hz and 0.32 mJ/mm2 , twice per week for 3 weeks
  Interventions: Device: Focused Extracorporeal Shock Wave Therapy (ESWT)
- Physiotherapy (Active Comparator): therapeutic ultrasound, 12 times in 3 weeks
  Interventions: Device: physiotherapy

INTERVENTIONS:
Device: Focused Extracorporeal Shock Wave Therapy (ESWT) — 2000 impulses of 5 Hz and 0.32 mJ/mm2 , twice per week for 3 weeks
  Arms: Focused Extracorporeal Shock Wave Therapy (ESWT)
Device: physiotherapy — therapeutic ultrasound, 12 times in 3 weeks
  Arms: Physiotherapy

SUMMARY:
Trigger finger is the common name of stenosing tenosynovitis of fingers, caused by repetitive trauma. Conservative treatment includes NSAIDs or other analgesic agents, activity modification, splint, and physiotherapy. Operation could be considered if conservative treatments fails. With literature reviewed, there is no treatment which is both non-invasive and effective, and also could avoid recurrence well.

Extracorporeal shock wave therapy could induce angiogenesis, anti-inflammatory reaction, and recruitment of fibroblast. Although extracorporeal shock wave has been utilized in musculoskeletal diseases for more than twenty years, there is no well-designed clinical trial to prove the effectiveness of extracorporeal shock wave in treating trigger finger. The purpose of this study is to compare the effectiveness of extracorporeal shock wave therapy with traditional physical therapy for the management of trigger finger.

ELIGIBILITY:
Inclusion Criteria:

* Quinnel classification grade 2 or 3
* who has only one trigger

Exclusion Criteria:

* who had ever treated the trigger finger
* who has other musculoskeletal disease of the upper limb
* who has severe coagulopathy disease
* who is pregnant
* who has arrhythmia or has a pacemaker
* there is sensory impairment, scar, edema at the trigger finger
* who has cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Quinnell stages of triggering | 15 weeks
  Quinnell stages of triggering classifies the trigger finger using five types during flexion and extension: normal movement (Type 0), uneven movement (Type I), actively correctable (Type II), passively correctable (Type III) and fixed deformity (Type IV).
11-point numeric scale of pain | 15 weeks
  The 11-point numeric scale of pain requires the patient to rate their pain on a defined scale. 0 is no pain and 10 is the worst pain imaginable.
Chinese quick DASH (disabilities of the Arm, Shoulder, and Hand questionnaire) | 15 weeks
  This questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The investigators chose the first two components: the disability and symptom section (11 items, scored 1-5). The lower score means better condition of upper limbs, and vice versa.
strength of hand grip | 15 weeks
  The strength of hand grip is to measure the maximum isometric strength of the hand and forearm muscles by a electicial grip strength device.
sonographic image | 15 weeks
  The investigators would record the characteristics of acquired sonographic images, such like the thickness of finger flexor tendon and A1 pulley, the presence of tendon sheath effusion, and the presence of increased vascularity by Doppler images.